CLINICAL TRIAL: NCT01799057
Title: Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Study of Metformin for the Assessment of Changes in Functional Capacity, Endothelial Function, and Hemodynamics in Individuals With Peripheral Artery Disease-Related Intermittent Claudication
Brief Title: The Effects of Metformin on Functional Capacity in Individuals With Peripheral Artery Disease-Related Intermittent Claudication
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial has been terminated due to difficulties with recruitment.
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 493/12
Record Dates: First submitted 2013-02-22; First posted 2013-02-26 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
Keywords: Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases; Vascular Diseases; Cardiovascular Diseases; Arterial Occlusive Diseases; Atherosclerosis; Insulin Resistance; Glucose Metabolism; Blood Glucose; Metformin; Biguanides; Hypoglycemic Agents; Endothelium, Vascular; Hemorheology; Blood Circulation; Regional Blood Flow; Microcirculation; Exercise; Physical Fitness; Exercise Test; Sedentary Lifestyle; Quality of Life; Plethysmography
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication; Peripheral Vascular Diseases; Vascular Diseases; Cardiovascular Diseases; Arterial Occlusive Diseases; Atherosclerosis; Insulin Resistance; Motor Activity; Sedentary Behavior | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin at a maximum dose of 1000mg twice daily for 16-18 weeks (i.e. maximum of 2000mg per day).
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Matching placebo twice daily for 16-18 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Participants randomized to metformin will be treated at a maximum dose of 2000mg per day (i.e. 1000mg twice daily for 16-18 weeks; up-titrated from 500mg twice daily for the first 2 weeks). Participants may complete the 16-18 week treatment intervention at the lower dose of 500mg twice daily if limited by side effects.
  Other Names: Diaformin
  Arms: Metformin
Drug: Placebo — Participants randomized to placebo will take matching oral capsules according to the same dose schedule specified for the metformin intervention.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of metformin on functional capacity (pain-free and maximum walking times) in individuals with peripheral artery disease (PAD)-related intermittent claudication.

DETAILED DESCRIPTION:
Background and Rationale:

Metformin has demonstrable efficacy in slowing or reversing the progression of various insulin-resistant disease states - most notably type 2 diabetes and pre-diabetes. In seeking to establish proof-of-concept that insulin resistance is a suitable pathophysiological target in the treatment of PAD-related intermittent claudication (pain in the leg muscles during walking, which resolves on exercise cessation), this study will determine whether the known insulin-sensitizing effects of metformin translate to alleviation of the functional limitations imposed by claudication.

Study Design:

A total of 80 individuals with PAD-related intermittent claudication will be randomised (1:1) to either metformin or matching placebo for 16-18 weeks (double-blind, parallel group design). The maximum daily dose of metformin will be 2000mg (up-titrated from half this dose at 2 weeks if tolerated).

Primary Hypothesis:

Improvement in functional capacity follows metformin therapy in individuals with PAD-related intermittent claudication. Change in functional capacity will be assessed by the co-primary endpoints of pain-free and maximum walking times during a standard graded treadmill exercise test.

Secondary Aims:

Exercise testing for functional performance will be complemented by assessments of perceived physical functioning / quality of life in the daily life setting (using standard questionnaires). As previous studies have indicated cardiovascular effects of metformin incremental to blood glucose-lowering, this study will also investigate potential mechanisms of efficacy relating to the primary endpoints, including changes in endothelial function, blood flow responses to various stimuli (including insulin and acute exercise), insulin sensitivity, and physical activity / sedentary behaviours. Changes in relevant clinical data (including ankle-brachial index and limb hemodynamics by duplex scanning) will also be determined.

Outcomes and Significance:

The unmet clinical need of efficacious medical therapies for intermittent claudication is a growing problem given the increasing prevalence of PAD worldwide. If positive, this study will identify a new potential treatment that is already widely available. The study will also inform on novel mechanistic targets with relevance to existing and future therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years old.
* Resting ankle-brachial index (ABI) ≤0.90 in the limiting leg(s), or a >20% reduction in the ABI measured immediately post-exercise where the resting ABI is >0.90. In cases of incompressible arteries in the limiting leg(s) (i.e. ABI ≥1.40), a toe-brachial index (TBI) of ≤0.70 is required.
* Peripheral artery stenosis/occlusion in the limiting leg(s), documented by duplex ultrasonography or other imaging tests.
* Stable (i.e. 3-month history) intermittent claudication in at least one PAD-affected leg.
* Maximum walking time during graded treadmill exercise testing (Gardner-Skinner protocol) ≥1 minute and ≤16 minutes.
* Concurrent medications that may affect primary, secondary or exploratory endpoints have remained stable over the previous 3 months.
* Have given signed informed consent to participate in the study.

Exclusion Criteria:

* Identification of any other medical condition requiring immediate therapeutic intervention.
* Clinically significant abnormal electrocardiogram (ECG) at rest or during exercise that represents a contraindication to study procedures or the study drug.
* Myocardial infarction, unstable angina, percutaneous transluminal coronary angioplasty (PTCA), coronary artery bypass graft surgery (CABG), or other major surgery within the previous 6 months.
* Exercise capacity limited by a factor other than PAD-related intermittent claudication.
* Any condition that precludes valid completion of a treadmill exercise test.
* Critical limb ischemia in either leg, defined as PAD-related chronic ischemic rest pain or skin lesions (ulcers, gangrene).
* Previous peripheral revascularisation or other surgical treatment for PAD in the previous 6 months.
* Known non-atherosclerotic cause of PAD.
* Active cancer.
* Uncontrolled hypertension (resting brachial blood pressure ≥160/100 mmHg).
* Evidence of pharmacologically-treated or poorly controlled (i.e. HbA1c ≥7.5%) type 2 diabetes or other class of diabetes (e.g. type 1 diabetes).
* Known intolerance or contraindication(s) to metformin.
* Known contraindication(s) to "Definity" (perflutren lipid microsphere).
* Participation or intention to participate in another clinical research study during the study period.
* History of non-compliance to medical regimens or unwillingness to comply with the study protocol.
* Any other condition that in the opinion of the Investigators would confound the evaluation and interpretation of the data.
* Persons directly involved in the execution of the protocol.
* Incapable of providing written informed consent due to cognitive, language, or other reasons.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in pain-free walking time | Measured at baseline and following 16-18 weeks treatment
  Pain-free walking time (time to onset of claudication) will be measured during a graded treadmill exercise test.
Change in maximum walking time | Measured at baseline and following 16-18 weeks treatment
  Maximum walking time will be measured during a graded treadmill exercise test.

SECONDARY OUTCOMES:
Change in questionnaire-based markers of quality of life / perceived functional capacity | Measured at baseline and following 16-18 weeks treatment
Change in endothelial function | Measured at baseline and following 16-18 weeks treatment
Change in skeletal muscle blood flow response to insulin | Measured at baseline and following 16-18 weeks treatment
Change in skeletal muscle blood flow response to acute exercise | Measured at baseline and following 16-18 weeks treatment
Change in insulin sensitivity | Measured at baseline and following 16-18 weeks treatment
Change in objectively measured physical activity / sedentary behaviour in the daily life setting. | Measured at baseline and following 16-18 weeks treatment

OTHER OUTCOMES:
Change in glucose uptake and insulin signalling mechanisms in skeletal muscle (exploratory endpoint) | Measured at baseline and following 16-18 weeks treatment
Change in skeletal muscle oxidative capacity and substrate utilization (exploratory endpoint) | Measured at baseline and following 16-18 weeks treatment
Change in inflammation, fibrinolysis and coagulation (exploratory endpoint) | Measured at baseline and following 16-18 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn A Kingwell, PhD, Principal Investigator — Baker Heart and Diabetes Institute; Stephen J Duffy, MD, PhD, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker IDI Heart and Diabetes Institute, Melbourne, Victoria, Australia